CLINICAL TRIAL: NCT03557164
Title: Intermediate and Long Term Vascular Effects of Cisplatin in Patients With Testicular Cancer
Acronym: INTELLECT
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: 16/WS/0030
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Testicular Cancer; Cardiovascular Diseases; Cardiovascular Risk Factor
MeSH Terms: conditions — Testicular Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chemotherapy drugs improve cancer survival but increase the risk of cardiovascular disease (CVD). VEGF inhibitors (VEGFI) cause severe hypertension, while cisplatin appears pro-thrombotic. Hence while cancer survival may improve, this is at the risk of potentially severe CVD and associated morbidity. Mechanisms underlying the cardiovascular toxicities of VEGFI and cisplatin are unknown, but effects on vascular function may be important.

The INTELLECT study will phenotype the endothelial effects of VEGFI and cisplatin using a variety of methods.

DETAILED DESCRIPTION:
There remains an unmet need to identify a preventive treatment for patients with testicular cancer treated with platinum based chemotherapy to diminish the risk of subsequent cardiovascular events. A future randomised trial of statin therapy in these patients is under consideration and results from this study will inform its design.

The information gained from this pilot study will guide the development of interventional pharmacological studies that are directed towards the most appropriate pathophysiological processes, at the most appropriate time and in the most appropriate patient groups treated with platinum based chemotherapy for testicular cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of stage 1 low-risk germ cell testicular cancer treated with orchidectomy, or IGCCC good or intermediate prognosis metastatic testicular/retroperitoneal germ cell cancer treated with orchidectomy (and or retroperitoneal surgery) plus cisplatin based chemotherapy, 12 - 18 months or 5 - 7 years previously.
* Aged between 18 and 50 years inclusive, at time of enrolment

Exclusion Criteria:

* Unable to provide written, informed consent
* Unable or unwilling to attend for investigations
* Current active involvement in a clinical trial
* Those receiving drug treatment for any vascular disease:

  o Including hypertension, hyperlipidaemia, cerebrovascular disease, ischaemic heart disease or heart failure
* Asthma
* Chronic obstructive pulmonary disease
* Diabetes mellitus
* Arial fibrillation/flutter
* Oral anticoagulation therapy
* Cigarette smoker or tobacco use
* Recreational drug use
* Ongoing inflammatory, infective or autoimmune disease
* Other malignant disease diagnosed in previous 7 years
* Previous venous or arterial thrombotic/thromboembolic event

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: testicular cancer oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
venous occlusion plethysmography assessment of endothelial function | 8 weeks
  expressed as ml per 100 ml of forearm volume per minute

CONTACTS AND LOCATIONS:
Overall Officials: Ninian Lang, MBChB PhD, Principal Investigator — QEUH, NHS Greater Glasgow and Clyde
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cameron AC, McMahon K, Hall M, Neves KB, Rios FJ, Montezano AC, Welsh P, Waterston A, White J, Mark PB, Touyz RM, Lang NN. Comprehensive Characterization of the Vascular Effects of Cisplatin-Based Chemotherapy in Patients With Testicular Cancer. JACC CardioOncol. 2020 Sep;2(3):443-455. doi: 10.1016/j.jaccao.2020.06.004. PMID 33043304